CLINICAL TRIAL: NCT00334555
Title: Control of Trichomoniasis - A Paradigm for STD Control
Brief Title: Control of Trichomoniasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Jane Schwebke, MD, University of Alabama at Birmingham
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: F020508005; R01AI050718 (NIH)
Record Dates: First submitted 2006-06-07; First posted 2006-06-08 (Estimated); Last update posted 2009-08-12 (Estimated); Status verified 2009-08

CONDITIONS: Trichomoniasis
Keywords: trichomoniasis; partner notification
MeSH Terms: conditions — Trichomonas Infections

ARMS (3):
- usual care (Active Comparator): patient told to refer her partner for treatment
  Interventions: Other: different methods of partner notification; Other: partner delivered meds; Other: field intervention
- partner delivered (Active Comparator): patient given medication to deliver to her partners
  Interventions: Other: partner delivered meds; Other: field intervention
- field intervention (Active Comparator): field intervention to find partners
  Interventions: Other: field intervention

INTERVENTIONS:
Other: different methods of partner notification — comparing patient referral, partner delivered medications and field intervention to treat sex partners
  Arms: usual care
Other: partner delivered meds — patient given meds to give to her partner
  Arms: partner delivered; usual care
Other: field intervention — health worker finds partners

SUMMARY:
This study is designed to try to find the best method of partner notification and treatment for partners of women with trichomonas

DETAILED DESCRIPTION:
To carry out a randomized trial to compare the effectiveness of three methods of partner notification and treatment for sexual partners of women with vaginal trichomoniasis - patient self-referral of partners (the current practice standard), delivery of curative therapy to partners by patients themselves, or public health style Disease Intervention carried out by a specially trained Disease Intervention Specialists (DIS) locating the partners and delivering the medication in the field. Reinfection rates with trichomonas at three months of follow-up among the index women will be the measure of effectiveness.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria {for Women}:

Age {> 15 years} Culture or wet prep proven T. vaginalis infection Willingness to provide informed consent and take part in study procedures

-

Exclusion Criteria:

* Exclusion criteria:

Infection with other STD pathogens requiring Health Dept DIS intervention (syphilis or HIV) Pregnancy or currently breast feeding Recent (8 hours) ingestion of alcoholic beverages or intent to do so in the 24 hours following treatment Allergy to metronidazole The presence of a sexual partner in the clinic at the time of enrollment A history of referral by a partner already treated for trichomoniasis Report of more than four sexual partners in the preceding 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 599 (Actual)
Dates: Start 2003-05; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
recurrence of trichomonas in the index patient | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jane Schwebke, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Jefferson County Department of Health STD Clinic, Birmingham, Alabama, United States